CLINICAL TRIAL: NCT03696147
Title: Role of Diffusion Magnetic Resonance Imaging in Assessment of Mammographically Detected Asymmetric Densities
Brief Title: Diffusion Magnetic Resonance Imaging in Mamographically Detected Asymmetric Densities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Ali Saad, Assistant lecturer, Assiut University
Other Study IDs: DWI breast cancer
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Mammographic Density
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Magnetic resonance imaging — Diffusion weighted sequence of MRI

SUMMARY:
The aim of the study is to identify the role of diffusion weighted MRI in the assessment of the clinical significance and outcomes of asymmetric breast densities identified on mammograms, and to identify the inconclusive mammographic findings most frequently associated with occult breast carcinoma.

DETAILED DESCRIPTION:
Although there is clearly a wide variation in breast size and parenchymal pattern, the breasts are generally symmetric structures with similar density and architecture. However, asymmetric breast tissue is encountered relatively frequently.

Asymmetric breast tissue is usually benign and secondary to variations in normal breast tissue, postoperative change from a previous biopsy, hormone replacement therapy , or merely poor positioning. However, an asymmetric area may indicate a developing mass or an underlying cancer.

The American College of Radiology (ACR), Breast Imaging Reporting and Data System (BI-RADS) defined four different types of asymmetric breast findings:

1. Asymmetric Breast tissue: refers to a greater volume or density of breast tissue in one breast than in the corresponding area in the contra lateral breast.
2. Densities seen in one projection: reflect a density seen in only one mammographic projection.
3. Architectural distortion: refers to a focal area of breast tissue that appears distorted with no definable central mass. Speculations radiate from a common point, and there is an area of focal retraction and tethering of normal parenchyma.
4. Focal asymmetric densities: refer to focal asymmetric densities that are seen on two mammographic views but cannot be accurately identified as a true mass.

These lesions are frequently encountered at screening and diagnostic mammography and are significant because they may indicate a neoplasm, especially if an associated palpable mass is present. Once these lesions are detected at standard mammography, supplementary breast imaging with additional mammographic views and ultrasonography (US) can be a key aspect of work-up.

However, these techniques may be insufficient to make a final BI-RADS assessment and may have limited sensitivity and specificity for the detection and diagnosis of breast lesions, yielding equivocal results. Certainty of the presence or absence of a true lesion can be difficult, and the findings remain inconclusive. Moreover, Architectural distortion should always be regarded with suspicion but differentiation from summation artifact is problematic. Developing asymmetric densities need to be evaluated unless they can be explained in terms of benign causes.

In these situations, MRI can be performed as an additional problem- solving procedure. Positive MRI examination will prompt biopsy and allow for the timely detection of malignancies that may otherwise would gone undiagnosed, while a negative MRI will allow increased confidence that the equivocal finding was likely caused by summation artifact or benign tissue , so follow-up surveillance mammography without biopsy will be undergone.

Although conventional breast MRI has a high sensitivity (89-100%) in the characterization of breast lesions . However, an overlap between benign and malignant findings still persists, resulting in a variable specificity (50-90%).

The DWI derives images from the difference of water molecules motion (Brownian motion) in tissues, resulting in quantitative and qualitative data reflecting changes at the cellular level and, consequently, unique information on the tumor cellularity and cell membranes integrity. This would allow the increase in breast MRI specificity and reduction of false-positive results and unnecessary biopsies.

Cell density might play an important role in the different ADCs obtained from benign and malignant breast lesions and the measurement of extracellular water content may be an additional feature that can improve MRI specificity.

The main objectives in using diffusion sequences are to optimize characterization of lesions differentiating benign from malignant tumors; and to improve detection of small lesions, which requires an optimal signal-to-noise ratio. several authors have shown that this technique is relevant for smaller masses (5 mm) and even for non-mass like enhancements.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented with asymmetric breast densities, seen on screening or diagnostic mammograms.

Exclusion Criteria:

* Patients with cardiac pacemakers.
* Patients with brain aneurysm clips.
* Patients with cochlear implants.
* Patients with vascular stents.
* Claustrophobic.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: sample size was calculated using EpiInfo7statcalc. Prog. With the following input population size: 120 expected frequency: 6% confidence limits: 5% design effect: 1.0 clusters: 1 The sample size was 50 cases at 95%confidence level.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of diffusion MRI finding with the pathology of the specimens | Baseline
  Analysis of diffusion weighted images and ADC values to defferntiate different pathologies causing asymmetric densities in routine screening or diagnostic mammography